CLINICAL TRIAL: NCT01745250
Title: A Randomised, Evaluator-blinded, Comparative Study of the Safety and Efficacy of Lip Injections With Emervel Lips and Juvederm Ultra Smile
Brief Title: Safety and Efficacy of Lip Injections With Emervel Lips and Juvederm Ultra Smile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05DF1210
Record Dates: First submitted 2012-12-04; First posted 2012-12-10 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2016-01

CONDITIONS: Local Tolerability After Lip Filler Injections
Keywords: lip; fillers; Hyaluronic acid
MeSH Terms: conditions — Lymphoid Interstitial Pneumonia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Emervel Lips (Experimental): Emervel Lips
  Interventions: Device: Emervel Lips
- Juvederm Ultra Smile (Experimental): Juvederm Ultra Smile
  Interventions: Device: Juvederm Ultra Smile

INTERVENTIONS:
Device: Emervel Lips — Lip treatment of both upper and lower lip
  Arms: Emervel Lips
Device: Juvederm Ultra Smile — Lip treatment of both upper and lower lip
  Arms: Juvederm Ultra Smile

SUMMARY:
The purpose of this study is to demonstrate the efficacy and safety of Emervel Lips and Juvederm Ultra smile

ELIGIBILITY:
Inclusion Criteria:

* Female subjects aged 18 to 65 years.
* Subjects with the intention to undergo lip augmentation treatment.
* Subjects treatment-naïve for lip augmentation treatment
* Subjects with lip appearance judged by the treating investigator to be suitable for lip line treatment
* Subjects with signed informed consent.

Exclusion Criteria:

* Concomitant anticoagulant therapy and therapy with inhibitors of platelet aggregation (e.g. aspirin or other nonsteroidal anti-inflammatory drugs [NSAIDs]), Omega-3 or vitamin E within 10 days before study treatment, or a history of bleeding disorders.
* Prior surgery or tattoo to the upper or lower lip or lip line.
* Presence of any abnormal lip structure, such as a scar or lump or severe lip asymmetry.
* Previous tissue augmenting therapy in the lip area (including oral commissures, marionette and perioral lines) with HA or collagen filler, or laser treatment, within 12 months before study entry.
* Permanent implant or treatment with non-HA or non-collagen filler in the area surrounding the lips (including nasolabial folds, oral commissures, marionette and perioral lines).
* History of herpes labialis with an outbreak within 4 weeks of study entry or with 4 or more outbreaks in the 12 months before study entry.
* Active skin disease, inflammation or related conditions, such as infection, psoriasis and herpes zoster near or on the area to be treated.
* History of angioedema.
* Previous hypersensitivity to HA.
* Previous hypersensitivity to lidocaine or other amide-type anaesthetics
* Cancerous or precancerous lesions in the area to be treated.
* Immunosuppressive therapy, chemotherapy, treatment with biologics or systemic corticosteroids within 3 months before study treatment.
* Pregnancy or breast feeding.
* Participation in any other clinical study within 30 days before inclusion.
* Other condition preventing the subject to entering the study in the investigator's opinion, e.g. subjects not likely to avoid other facial cosmetic treatments below the level of the lower orbital rim, subjects anticipated to be unreliable or incapable of understanding the study assessment or unrealistic expectations of treatment result.
* Study staff or close relative to study staff (e.g. parents, children, siblings or spouse).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Local tolerability | 14 days
  To assess local tolerability after treatment including erythema, bruising, itching, swelling, pain/ tenderness at 14 days. Number of subjects reporting the events will be analysed.

SECONDARY OUTCOMES:
AE reporting | 24 weeks
  To evaluate long-term safety throughout the study period
Global Aesthetic Improvement Scale (GAIS) | Week 2 to week 24
  To evaluate esthetic change of lips from baseline using GEIS
Lip Fullness Grading Scale (LFGS) | 0-24 weeks
  To evaluate esthetic change of lips from baseline using LFGS
Subject's satisfaction | 0-24 weeks
  To evaluate subjects satisfaction in terms of a subject satisfaction questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Said Hilton, MD, Principal Investigator — Medical Skin Center
Locations (1):
- Medical Skin center, Düsseldorf, Germany